CLINICAL TRIAL: NCT04516343
Title: Development of a Robotic Ankle Assist Device to Improve Mobility in Individuals With Movement Disorders
Brief Title: Development of a Robotic Ankle Assist Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BiOMOTUM, Inc. (Industry)
Collaborators: Northern Arizona University (Other); Gillette Children's Specialty Healthcare (Other); Shirley Ryan AbilityLab (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R44HD104328 (NIH)
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: This study has two experiments. In experiment I, participants will be recruited to complete gait training with the RAAD under assistance mode. In experiment two, participants will be recruited to complete gait training with the RAAD under resistance mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Therapist supervised assistance training (Experimental): Assistance training with the RAAD under therapist supervision.
  Interventions: Device: Robotic Ankle Assist Device (RAAD)
- Therapist supervised resistance training (Experimental): Resistance training with the RAAD under therapist supervision.
  Interventions: Device: Robotic Ankle Assist Device (RAAD)

INTERVENTIONS:
Device: Robotic Ankle Assist Device (RAAD) — The RAAD (Robotic Ankle Assist Device) is an intelligent, powered ankle device designed to increase independence, mobility, and deliver gait training to children with movement disorders, such as CP

SUMMARY:
The overall objectives of this work is to establish feasibility of a robotic ankle assist device (RAAD) to improve mobility in free-living settings and to establish the RAAD as an effective tool to provide increased dose and precision of targeted ankle therapy.

The first specific goal is to assess the benefits of repeated gait training with RAAD assistance. Individuals with CP will participate in a 4-week assistance intervention and mobility outcomes will be quantified pre and post intervention.

The second specific goal is to separately assess the benefits of repeated gait training with RAAD resistance. Individuals with CP will participate in a 4-week resistance intervention and mobility outcomes will be quantified pre and post intervention.

Assessed separately, it is hypothesized that both assistance and resistance training will improve mobility outcomes.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of cerebral palsy. Any sex, race, ethnicity or socioeconomic status. GMFCS level I, II, or II. Ability to walk for at least 6 minutes (assisted or unassisted). Age between 8-18 years. Height/weight/BMI between the 5th - 95th percentile of children with CP.

Able to understand and follow simple directions. Able to complete 5 heel raises with minimal assistance (balance only). At least 20 degrees of passive ankle plantar flexion range of motion.

Exclusion Criteria:

Knee extension or ankle dorsiflexion contractures greater than 15 degrees. Health condition or diagnosis other than CP that would affect safe participation.

Orthopedic surgery completed in the prior 12-months. Current enrollment in a conflicting research study.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray Browning, PhD, Principal Investigator — BiOMOTUM, Inc.
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Therapist Supervised Assistance Training: One group of participants were recruited to complete assistance training with the RAAD under therapist supervision.
  Robotic Ankle Assist Device (RAAD): The RAAD (Robotic Ankle Assist Device) is an intelligent, powered ankle device designed to increase independence, mobility, and deliver gait training to children with movement disorders, such as CP
- Therapist Supervised Resistance Training: A second group of participants were recruited to complete resistance training with the RAAD under therapist supervision.
  Robotic Ankle Assist Device (RAAD): The RAAD (Robotic Ankle Assist Device) is an intelligent, powered ankle device designed to increase independence, mobility, and deliver gait training to children with movement disorders, such as CP
Period: Overall Study
Arm/Group | Therapist Supervised Assistance Training | Therapist Supervised Resistance Training
Started | 12 | 19
Completed | 12 | 16
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapist Supervised Assistance Training | Therapist Supervised Resistance Training | Total
Number analyzed (Participants) | 12 | 19 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.6 (3.3) | 13.2 (3.9) | 13.4 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 6 | 11 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 11
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 7
Region of Enrollment [Number; unit: participants]
  United States | 12 | 19 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Preferred Walking Speed
Description: How fast someone prefers to walk
Time Frame: baseline and post intervention at 6 minutes
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Therapist Supervised Assistance Training | Therapist Supervised Resistance Training
Number analyzed (Participants) | 12 | 16
m/s | 0.09 (0.13) | 0.13 (0.14)

2. Secondary Outcome: Change in COT
Description: Change in Metabolic cost of transport
Time Frame: baseline and post intervention
Population: 6 participants were unable to complete this outcomes measure test because of the metabolic face mask.
Measure: Mean (Standard Deviation); unit: J/kg/m
Arm/Group | Therapist Supervised Assistance Training | Therapist Supervised Resistance Training
Number analyzed (Participants) | 12 | 10
J/kg/m | -0.06 (0.13) | -0.01 (0.11)

3. Secondary Outcome: Change in 6MWT
Description: Change in Six-minute walk test, which is the total distance walked over a 6 minute period.
Time Frame: 6 minutes pre/post
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Therapist Supervised Assistance Training | Therapist Supervised Resistance Training
Number analyzed (Participants) | 12 | 16
m | 46 (53.7) | 48.4 (74.2)

4. Secondary Outcome: Change in Gait Kinetics
Description: Change in Average knee angle across stance phase measured in degrees
Time Frame: 6 minutes pre/post
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Therapist Supervised Assistance Training | Therapist Supervised Resistance Training
Number analyzed (Participants) | 11 | 12
degrees | -1.62 (2.05) | -2.00 (6.89)

5. Secondary Outcome: Change in Step Length
Description: Step length during walking
Time Frame: baseline and post intervention
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Therapist Supervised Assistance Training | Therapist Supervised Resistance Training
Number analyzed (Participants) | 11 | 13
m | 0.082 (0.184) | 0.072 (0.142)

6. Secondary Outcome: Change in Gross Motor Function Measure Scale 66
Description: Change in Gross motor function measure scale 66, min score = 0, max score = 66, high score is better. Unit of measure = Scores on a scale.
Time Frame: 20 minutes pre/post
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Therapist Supervised Assistance Training | Therapist Supervised Resistance Training
Number analyzed (Participants) | 12 | 16
scores on a scale | 1.43 (3.1) | 1.56 (2.032)

7. Secondary Outcome: Change in Fast Walking Speed
Description: How fast participants prefer to walk quickly (m/s)
Time Frame: baseline and post intervention
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Therapist Supervised Assistance Training | Therapist Supervised Resistance Training
Number analyzed (Participants) | 12 | 14
m/s | 0.06 (0.18) | 0.18 (0.21)

ADVERSE EVENTS:
Time Frame: During the protocol, approximately 4 weeks
Arm/Group | Therapist Supervised Assistance Training | Therapist Supervised Resistance Training
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/16
Other Adverse Events (participants affected / at risk) | 3/12 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapist Supervised Assistance Training (N=12) | Therapist Supervised Resistance Training (N=16)
Fall (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — A fall during the walking protocol

LIMITATIONS AND CAVEATS:
Some participants were unable to complete all assessment tests leading to small sample sizes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT04516343/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT04516343/SAP_001.pdf
  • Informed Consent Form (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT04516343/ICF_002.pdf